CLINICAL TRIAL: NCT01488903
Title: A Cohort Research of Genetic Susceptibility for Common Obesity in Women (CROWN Study)
Brief Title: A Cohort Research of Genetic Susceptibility for Common Obesity in Women
Acronym: CROWN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, vghtpe user, Principal Investgator, Taipei Veterans General Hospital, Taiwan
Other Study IDs: 2011-06-013GA
Record Dates: First submitted 2011-12-06; First posted 2011-12-08 (Estimated); Last update posted 2011-12-14 (Estimated); Status verified 2011-12

CONDITIONS: Obesity; Menopause
Keywords: genetic susceptibility; obesity; body composition; the metabolic syndrome; women
MeSH Terms: conditions — Obesity; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA, fasting blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Premenopausal Women: 600 health premenopausal Women
- Postmenopausal women: 600 healthy postmenopausal women

SUMMARY:
Not many studies examined genetic determinants of obesity in women. As pre-menopausal and post-menopausal women appear to have different propensities for fat deposition, genetic loci linked with obesity-related phenotypes might be different by menopausal status. So far, there is no large scale of genetic study deciphering common obesity focusing on women population to examine the contributions of aging and change in menopausal status to obesity in Taiwan. The investigators propose this study to compare phenotypic profiles of obesity and cardio-metabolic factors in pre-menopausal and post-menopausal women. The study will examine the contributions of aging and change in menopausal status to the changes of obesity-related traits during the transition from pre-menopause to post-menopause period, and will evaluate the contribution of genetic susceptibility on body fat deposition among women at different stage of menopause.

DETAILED DESCRIPTION:
Not many studies examined genetic determinants of obesity in women. As premenopausal and postmenopausal women appear to have different propensities for fat deposition, genetic loci linked with obesity-related phenotypes might be different by menopausal status. So far, there is no large scale of genetic study deciphering common obesity on women focusing on the interaction between aging and menopause in Taiwan. The investigators propose this study to compare phenotypic profiles of obesity and cardiometabolic factors in a large group of premenopausal and postmenopausal women. The study will examine the contributions of aging and menopausal status to the changes of obesity-related traits, and will evaluate the contribution of genetic susceptibility on body fat deposition among women at different stage of menopause. The investigators plan to recruit two groups of subjects: 600 premenopausal, and 600 postmenopausal women. Each woman will receive anthropometric and blood pressure measurements, fasting blood sampling for lipids, and an optional 75-g oral glucose tolerance test for insulin resistance. Dual energy X-ray absorptiometry will also be used for body composition measurements among the study women if they agree to receive this optional examination. The investigators will collect blood samples for DNA extraction and select several candidate genes to study the associations between susceptible genes and obesity-related traits. The investigators anticipate that the results generated from the study will provide valuable data to a better understanding of the pathogenesis of common obesity during transition from premenopause to postmenopause in women.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal Women Group
* Age: 35 ~ 50 years old
* Subjects have menstrual period
* Subjects are not pregnant
* Subject is willing to sign inform consent
* Postmenopausal Women Group
* Age: 50 ~ 65 years old
* Women who have not menstruated within the last 12 months
* Subject is willing to sign inform consent.

Exclusion Criteria:

* Pregnant women
* Women with known diabetes and fasting plasma glucose (PG) higher than 126 mg/dL
* Women have liver, kidney, heart and neurological diseases, as well as they have history of hyper- and hypothyroidism
* Subject has acute illness in the past 6 months
* Subject has history of alcohol or substance abuse
* Taking concomitant medication including hormone replacement and anti-lipid agents in two weeks
* Women with difficult giving venous blood sample

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The design of the project is a hospital-based case-control study. We will recruit two study groups: 600 post-menopausal women; 600 premenopausal women.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2011-09; Primary Completion 2014-07 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
genetic associations with body-mass index and waist circumference. | 3 years
  genetic associations with body-mass index and waist circumference.

SECONDARY OUTCOMES:
genetic associations with body fat composition | 3 years
  genetic associations with body fat composition, measured by DEXA
genetic associations with the metabolic syndrome | 3 years
  genetic associations with the metabolic syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Chii-Min Hwu, MD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan